CLINICAL TRIAL: NCT06010004
Title: A Phase 3, Long-term Safety Study of LY3502970 in Adult Participants With Type 2 Diabetes and Inadequate Glycemic Control With Diet and Exercise Alone or in Combination With Oral Antihyperglycemic Medications (ACHIEVE-J)
Brief Title: A Long-term Safety Study of Orforglipron (LY3502970) in Participants With Type 2 Diabetes
Acronym: ACHIEVE-J
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18745; J2A-JE-GZPE (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-08-21; First posted 2023-08-24 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — orforglipron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Orforglipron Dose 1 (Experimental): Participants will receive orforglipron administered orally.
  Interventions: Drug: Orforglipron
- Orforglipron Dose 2 (Experimental): Participants will receive orforglipron administered orally.
  Interventions: Drug: Orforglipron
- Orforglipron Dose 3 (Experimental): Participants will receive orforglipron administered orally.
  Interventions: Drug: Orforglipron

INTERVENTIONS:
Drug: Orforglipron — Administered orally
  Other Names: LY3502970

SUMMARY:
The purpose of this study is to determine the long-term safety of the study intervention orforglipron as a monotherapy or in combination with oral antihyperglycemic medication.

This study includes 3 periods as follows:

* screening and lead-in period: up to 4 weeks
* treatment period: 52 weeks, including 20 weeks of dose escalation, and
* safety follow-up period: 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have Type 2 Diabetes (T2D)
* Have HbA1c ≥7.0% (≥53 mmol/mol) to ≤10.5% (≤91 mmol/mol) as determined by the central laboratory at screening.
* Are of stable weight (±5%) for at least 90 days prior to screening and agree to not initiate an intensive diet or exercise program during the study with the intent of reducing body weight other than the lifestyle and/or dietary measures for diabetes treatment.
* Have a BMI ≥23.0 kilogram/square meter (kg/m²) at screening.

Exclusion Criteria:

* Have Type 1 Diabetes (T1D).
* Have a history of severe hypoglycemia or hypoglycemia unawareness within the last 6 months prior to screening, or between screening and randomization.
* Have New York Heart Association functional classification IV congestive heart failure.
* Have had any of the following cardiovascular (CV) conditions within 60 days prior to screening, or between screening and randomization.

  * acute myocardial infarction
  * cerebrovascular accident (stroke), or
  * hospitalization for congestive heart failure
* Have acute or chronic hepatitis and pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Actual)
Dates: Start 2023-09-28 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | Baseline through Week 52

SECONDARY OUTCOMES:
Change from Baseline in Hemoglobin A1c (HbA1c) | Baseline, Week 52
Percentage of Participants who Achieve HbA1c <7.0% (<53 mmol/mol) | Week 52
Percentage of Participants who Achieve HbA1c ≤6.5% (<48 mmol/mol) | Week 52
Percentage of Participants who Achieve HbA1c <5.7% (<39 mmol/mol) | Week 52
Change from Baseline in Fasting Serum Glucose | Baseline, Week 52
Change from Baseline in Body Weight | Baseline, Week 52
Percentage of Participants who Achieve Weight Loss of ≥5% | Week 52
Percentage of Participants who Achieve Weight Loss of ≥10% | Week 52
Percentage of Participants who Achieve Weight Loss of ≥15% | Week 52
Change from Baseline in Waist Circumference | Baseline, Week 52
Change from Baseline in Body Mass Index (BMI) | Baseline, Week 52
Change from Baseline in Daily Average 7-Point Self-Monitored Blood Glucose (SMBG) | Baseline, Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (40):
- Japan (40):
  - Nakayama Clinic, Nagoya, Aichi-ken
  - Shinkashiwa Clinic, Kashiwa, Chiba
  - Kashiwa City Hospital, Kashiwa, Chiba
  - Tokuyama Clinic, Mihama-ku,Chiba City, Chiba
  - Mikannohana Clinic, Diabetes, Endocrinology and Metabolism, Matsuyama, Ehime
  - Steel Memorial Yawata Hospital, Kitakyushu, Fukuoka
  - Hasegawa Medical Clinic, Chitose, Hokkaido
  - Odori Diabetes, Sapporo, Hokkaido
  - Matsuda Clinic, Kobe, Hyōgo
  - Nakamoto Internal Medicine Clinic, Mito, Ibaraki
  - MinamiAkatsukaClinic, Mito, Ibaraki
  - Nakakinen clinic, Naka, Ibaraki
  - Nishiyamadou Keiwa Hospital, Naka, Ibaraki
  - Taya Clinic Koueikai Medical Corporation, Tsuchiura, Ibaraki
  - Shonan Takai Clinic, Kamakura, Kanagawa
  - Takai Internal Medicine Clinic, Kamakura-shi, Kanagawa
  - Medical Corporation Yuga Tsuruma Kaneshiro Diabetes Clinic, Yamato-shi, Kanagawa
  - Yokohama Minoru Clinic, Yokohama, Kanagawa
  - Yokkaichi Diabetes Clinic, Yokkaichi, Mie-ken
  - Gibo Hepatology Clinic, Matsumoto, Nagano
  - Shiraiwa Medical Clinic, Kashihara, Osaka
  - Kitada Clinic, Osaka, Osaka
  - Medical Corporation Heishinkai OCROM Clinic, Suita-shi, Osaka
  - OHAMA Diabetes Clinic, Kawaguchi, Saitama
  - Sugiura Internal Medicine Clinic, Sōka, Saitama
  - Seiwa Clinic, Adachi-ku, Tokyo
  - The Institute for Adult Disease, Asahi Life Foundation, Chuo-ku, Tokyo
  - Tokyo-Eki Center-building Clinic, Chuo-ku, Tokyo
  - Fukuwa Clinic, Chuo-ku, Tokyo
  - Hachioji Diabetes Clinic, Hachioji-shi, Tokyo
  - Kanno Naika, Mitaka, Tokyo
  - Heishinkai Medical Group ToCROM Clinic, Shinjuku-ku, Tokyo
  - Medical Corporation Tao Internal Medicine Clinic, Ube, Yamaguchi
  - Fujii Clinic, Ube, Yamaguchi
  - Tashiro Endocrinology Clinic, Fukuoka
  - Morinaga Ueno Clinic, Kumamoto
  - Jinnouchi Hospital, Kumamoto
  - Heiwadai Hospital, Miyazaki
  - Kansai Electric Power Hospital, Osaka
  - Abe Clinic, Ōita

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Phase 3, Long-term Safety Study of LY3502970 in Adult Participants With Type 2 Diabetes and Inadequate Glycemic Control With Diet and Exercise Alone or in Combination With Oral Antihyperglycemic Medications (ACHIEVE-J) — https://trials.lilly.com/en-US/trial/419717